CLINICAL TRIAL: NCT07013643
Title: An Open-label, Single-sequence Multiple Cohort Study to Assess the Effect of Multiple Doses of AZD6234 and a Combination of AZD9550 and AZD6234 on the Pharmacokinetics of Single Doses of Combined Oral Contraceptive Ethinyl Estradiol/Levonorgestrel in Healthy Female Participants Living With Overweight or Obesity
Brief Title: A Study to Investigate the Effect of AZD6234 and a Combination of AZD9550 and AZD6234 on Pharmacokinetics of Combined Oral Contraceptive Ethinyl Estradiol/Levonorgestrel in Healthy Female Participants Living With Overweight or Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8750C00006
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Obesity; Overweight; Oral contraceptives; Pharmacokinetics; Drug Interaction
MeSH Terms: conditions — Obesity; Overweight | interventions — Ethinyl Estradiol; Levonorgestrel; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort-1 AZD6234 + EE/LEVO + Acetaminophen (APAP) (Experimental): Participants will receive combined oral contraceptive (EE/LEVO) and, separately, APAP, treatments throughout the study during the up-titration and maintenance periods of subcutaneous AZD6234 administration.
  Interventions: Drug: AZD6234; Drug: Ethinyl estradiol/Levonorgestrel (EE/LEVO); Drug: Acetaminophen (APAP)
- Cohort-2: AZD6234+AZD9550+EE/LEVO+APAP (Experimental): All participants will receive combined oral contraceptive EE/LEVO and separately, APAP, treatments throughout the study during the up-titration and maintenance periods of subcutaneous administered AZD6234 and AZD9550.
  Interventions: Drug: AZD6234; Drug: Ethinyl estradiol/Levonorgestrel (EE/LEVO); Drug: Acetaminophen (APAP); Drug: AZD9550

INTERVENTIONS:
Drug: AZD6234 — AZD6234 will be administered as a subcutaneous injection in the abdomen.
Drug: Ethinyl estradiol/Levonorgestrel (EE/LEVO) — EE/LEVO will be administered as combined oral tablets.
Drug: Acetaminophen (APAP) — APAP will be administered orally as a solution.
Drug: AZD9550 — AZD9550 will be administered as a subcutaneous injection in the abdomen.
  Arms: Cohort-2: AZD6234+AZD9550+EE/LEVO+APAP

SUMMARY:
This study will measure the effects of multiple doses of AZD6234 and a combination of AZD6234 and AZD9550 given as injection(s) on pharmacokinetics (PK) of combined oral contraceptive ethinyl estradiol (EE)/levonorgestrel (LEVO) in healthy female participants with obesity.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single-sequence, multiple-cohort study which will be performed at multiple study sites in healthy females of childbearing and non-childbearing potential.

The purpose of this study is to investigate the effect of AZD6234 and a combination of AZD6234 and AZD9550 on the PK, safety and tolerability of a combined oral contraceptive, ethinyl estradiol/levonorgestrel (EE/LEVO).

The study will have 2 cohorts, and each cohort will consist of 5 periods which include, Screening, Start, Up-titration, Maintenance, and Follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and if heterosexually active, must agree to use an approved method of highly effective contraception.

  o Hormonal contraceptives and estrogen-containing hormonal methods of birth control are not permitted due to potential effect and influence on the results using a combined oral contraceptive assessment.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Have a Body Mass Index (BMI) ≥ 25 kg/m2 inclusive and weigh at least 60 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder (gastroparesis, deep vein thrombosis, venous thromboembolism, previous surgery of the upper gastrointestinal tract, cardiovascular disease, neuromuscular or neurogenic disease, severe vitamin D deficiency, type I or type II diabetes mellitus, glycated hemoglobin (HbA1c) ≥ 6.5% at screening, history of neoplastic disease, basal calcitonin level >50 ng/L (50 pg/L) at screening (Cohort 2), history of acute or chronic pancreatitis or pancreatic amylase or lipase >2×ULN at screening (cohort 2), prior history of cholecystectomy or untreated cholelithiasis and personal or family history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia type 2 (MEN2) (cohort 2)).
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma.
* Any laboratory values with deviations or clinically important abnormalities in clinical chemistry, hematology, or urinalysis.
* Any positive result on screening for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb) or Human immunodeficiency virus (HIV).
* Abnormal vital signs.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12 lead electrocardiogram (ECG), at screening.
* Current smokers or those who have smoked or used nicotine products.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Statin treatment within 4 weeks prior to the start of study treatment.
* Current use of estrogen-containing products.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUCinf) of EE and LEVO | Cohort 1: At predefined intervals from Day -5 up to Day 99; Cohort 2 : At pre-defined interval from Day -5 up to Day 169
  To assess the effect of multiple doses of AZD6234 and, multiple doses of co-administered AZD9550 and AZD6234 on the PK of single doses of combined oral contraceptive EE/LEVO.
Area under the concentration-time curve from time of dosing to the last measurable concentration (AUClast) of EE and LEVO | Cohort 1: At predefined intervals from Day -5 up to Day 99; Cohort 2: At pre-defined interval from Day -5 up to Day 169
  To assess the effect of multiple doses of AZD6234 and, multiple doses of co-administered AZD9550 and AZD6234 on the PK of single doses of combined oral contraceptive EE/LEVO.
Maximum plasma concentration (Cmax) of EE and LEVO | Cohort 1: At predefined intervals from Day -5 up to Day 99; Cohort 2: At pre-defined interval from Day -5 up to Day 169
  To assess the effect of multiple doses of AZD6234 and, multiple doses of co-administered AZD9550 and AZD6234 on the PK of single doses of combined oral contraceptive EE/LEVO.
Time to reach maximum drug concentration in plasma (tmax) of EE and LEVO | Cohort 1: At predefined intervals from Day -5 up to Day 99; Cohort 2: At pre-defined interval from Day -5 up to Day 169
  To assess the effect of multiple doses of AZD6234 and, multiple doses of co-administered AZD9550 and AZD6234 on the PK of single doses of combined oral contraceptive EE/LEVO.
Elimination half-life (t1/2λz) of EE and LEVO | Cohort 1: At predefined intervals from Day -5 up to Day 99; Cohort 2: At pre-defined interval from Day -5 up to Day 169
  To assess the effect of multiple doses of AZD6234 and, multiple doses of co-administered AZD9550 and AZD6234 on the PK of single doses of combined oral contraceptive EE/LEVO.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Cohort 1: Up to Day 120; Cohort 2: Up to Day 216
  To assess the safety and tolerability of AZD6234 and co-administered AZD9550 and AZD6234 with combined oral contraceptive EE/LEVO.
Number of participants developing detectable anti-drug antibodies (ADAs) against AZD6234 and AZD9550 | Cohort 1: At predefined intervals from Day -2 up to Day 120; Cohort 2: At predefined intervals from Day -2 up to Day 216
  To assess the safety and tolerability of AZD6234 and co-administered AZD9550 and AZD6234 with combined oral contraceptive EE/LEVO.
Area under plasma concentration-time curve from time 0 to 168 hours postdose (AUC0-168h) of AZD6234 | Cohort 1: At predefined intervals from Day 1 to Day 120; Cohort 2: At predefined intervals from Day 8 to Day 216
  To characterize the PK of single and multiple doses of AZD6234 alone or in combination with AZD9550.
AUClast of AZD6234 | Cohort 1: At predefined intervals from Day 1 to Day 120; Cohort 2: At predefined intervals from Day 8 to Day 216.
  To characterize the PK of single and multiple doses of AZD6234 alone or in combination with AZD9550.
Cmax of AZD6234 | Cohort 1: At predefined intervals from Day 1 to Day 120; Cohort 2: At predefined intervals from Day 8 to Day 216
  To characterize the PK of single and multiple doses of AZD6234 alone or in combination with AZD9550.
AUC0-168h of AZD9550 | Cohort 1: At predefined intervals from Day 1 to Day 120; Cohort 2: At predefined intervals from Day 8 to Day 216
  To characterize the PK of single and multiple doses of AZD6234 alone or in combination with AZD9550.
AUClast of AZD9550 | Cohort 1: At predefined intervals from Day 1 to Day 120; Cohort 2: At predefined intervals from Day 8 to Day 216
  To characterize the PK of single and multiple doses of AZD6234 alone or in combination with AZD9550.
Cmax of AZD9550 | Cohort 1: At predefined intervals from Day 1 to Day 120; Cohort 2: At predefined intervals from Day 8 to Day 216
  To characterize the PK of single and multiple doses of AZD6234 alone or in combination with AZD9550.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/